CLINICAL TRIAL: NCT00465647
Title: A Multi-center, Open-label, Dose Titration Study Pharmacokinetics/Pharmacodynamics, Safety, and Efficacy of Hydromorphone Oral Solution in Subjects From 28 Days to 16 Years of Age, Who Require Opioid Analgesics for Postoperative Pain
Brief Title: An Open-label Study of Hydromorphone Oral Solution in Subjects Aged 28 Days to 16 Years for Postoperative Pain
Acronym: Palladone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMP4009
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Hydromorphone oral solution; opioid; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ≥ 28 Days to < 13 Months (Experimental): infant and toddler
  Interventions: Drug: Hydromorphone
- ≥ 13 months to < 5 years (Experimental): young child
  Interventions: Drug: Hydromorphone
- ≥ 5 years to < 12 years (Experimental): older child
  Interventions: Drug: Hydromorphone
- ≥ 12 years to < 17 years (Experimental): adolescent
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Oral hydromorphone solution dosed every 6 hours up to 9 doses. Dose is determined based on the expected weight range for each age group.
  Other Names: Infants and todlers;; Young child;; Older child;; Adolescent.

SUMMARY:
The primary objective of this study is to characterize the pharmacokinetics and pharmacodynamics of hydromorphone oral solution in pediatric subjects aged 28 days to 16 years inclusive. The secondary objectives are to characterize the safety and efficacy of hydromorphone oral solution in pediatric subjects aged 28 days to 16 years inclusive.

DETAILED DESCRIPTION:
Hydromorphone is an opioid analgesic that has been used for decades as an alternative to morphine in the treatment of moderate to severe malignant and nonmalignant pain. Only a small number of analgesics have been studied in children. The benefits to the subjects include contribution of knowledge that will provide for appropriate dosing regimen recommendations for future pediatric subjects.

Treatment consisted of both parenteral and oral hydromorphone. For up to 48 hours immediately following surgery, subjects were administered hydromorphone by IV PCA pump. Dosing with the oral hydromorphone HCl began when the subject was ready to take clear oral liquid. Subjects were administered oral hydromorphone HCl every 6 hours for up to 9 doses. The investigator determined the timing of the first dose based on each subject's clinical condition.

The duration of the treatment phase was up to 102 hours (up to 48 hours for the Parenteral Treatment Period and up to 54 hours for the Oral Treatment Period).

Efficacy was based on the oral hydromorphone treatment. Adverse events were collected for both the oral and parenteral treatments.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects aged 28 days to 16 years,
* Prospective subjects anticipated to have postoperative pain requiring oral opioid analgesics for at least 24 hours (up to 48 hours) following postoperative parenteral analgesia (up to 48 hours),
* Prospective subjects have received no more than a total of 7 doses of opioids in the 30 days prior to surgery.

Exclusion Criteria:

* Prospective subjects with clinically significant hepatic or renal dysfunction and impaired cardiac and/or respiratory reserve,
* Prospective subjects who have received opioid analgesic therapy other than hydromorphone or morphine sulfate during the up to 48-hour postoperative period prior to administration of first dose of oral hydromorphone,
* Prospective subjects who have received regional anesthetic blockade OR analgesic treatment with nonopioid medication within 6 hours prior to administration of first dose of oral hydromorphone.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 28 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory B. Hammer, MD, Principal Investigator — Stanford University
Locations (14):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County - Pediatric Subspecialty, Orange, California
  - Stanford University Medical Center, Stanford, California
  - The Children's Hospital, Aurora, Colorado
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Saint Louis University - Department of Neurology and Psychiatry, St Louis, Missouri
  - The University of North Carolina - CH, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Medical Center, Dallas, Texas
  - Texas Children's Hospital / Baylor College of Medicine, Houston, Texas
  - The University of Texas, Health Sciences Center at Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23-Apr-2007 (first subject, first visit) to 03-May-2009 (last subject, last visit). Multicenter study conducted at 18 sites in the United States (US).
Pre-assignment Details: Subjects who were anticipated to have acute, postoperative pain requiring oral opioid analgesics for at least 24 to 48 hours following postoperative parenteral analgesia.
Groups:
- ≥ 28 Days to < 13 Months: Infant and toddler - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- ≥ 13 Months to < 5 Years: Young child - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- ≥ 5 Years to <12 Years: Older child - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- ≥ 12 Years to < 17 Years: Adolescent- received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
Period: Overall Study
Arm/Group | ≥ 28 Days to < 13 Months | ≥ 13 Months to < 5 Years | ≥ 5 Years to <12 Years | ≥ 12 Years to < 17 Years
Started | 39 | 23 | 29 | 25
Completed | 26 | 15 | 18 | 12
Not Completed | 13 | 8 | 11 | 13
Not completed — Administrative | 2 | 2 | 3 | 2
Not completed — Adverse Event | 2 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 7
Not completed — The "other" reasons included loss of IV | 8 | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- ≥ 5 Years to < 12 Years: Older child - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- ≥ 12 Years to < 17 Years: Adolescent - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- Total: Total of all reporting groups
Arm/Group | ≥ 28 Days to < 13 Months | ≥ 13 Months to < 5 Years | ≥ 5 Years to < 12 Years | ≥ 12 Years to < 17 Years | Total
Number analyzed (Participants) | 39 | 23 | 29 | 25 | 116
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.9 (2.76) | 33.6 (14.90) | 105.9 (27.06) | 178.3 (17.05) | 73.5 (69.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 14 | 18 | 60
  Male | 21 | 13 | 15 | 7 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5 | 3 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 2 | 10 | 5 | 23
  White | 28 | 16 | 18 | 20 | 82
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Population Pharmacokinetic/Pharmacodynamic (PK/PD) Model for Hydromorphone: Clearance (Cl)
Description: Model was built using sparse blood samples: Sampling times: immediately predose, and between 0.25-0.75, 1-3, and 4-6 hours postdose for the first 2 doses of oral hydromorphone: predose for each dose of oral hydromorphone HCl thereafter; and at the end of study.
  Efficacy was based on Oral treatment only.
Time Frame: A maximum of 9 oral hydromorphone doses with potentially up to 54 hours duration.
Population: The full analysis population for Pharmacokinetics/ Pharmacodynamics consisted of subjects who received at least 1 dose of oral hydromorphone HCl, and had at least 1 valid quantifiable PK sample. To be a valid sample, the time of administration of each dose of oral hydromorphone HCl, the dose, and the time of sample collection must be recorded.
Measure: Number (95% Confidence Interval); unit: L/hour
Groups:
- All Patients: A total of all 4 age groups: infant and toddler, young child, older child, and adolescent.
Arm/Group | All Patients
Number analyzed (Participants) | 99
L/hour | 114 [80.6 to 203]

2. Secondary Outcome: Mean (SE) of Faces, Legs Activity, Cry, Consolability (FLACC) Pain Scores on Hydromorphone Alone (Oral/Supplemental) Over Time [Ages >=28 Days to <5 Years]
Description: There are 5 categories in this pediatric pain measurement: face, legs, activity, cry, and consolability. Responses in each category are scored between 0 and 2 (0 = normal, relaxed to 2 = upset, agitated), for a maximum total score of 10. The FLACC scale was used for children under the age of 3 years and older children who have limited verbal skills.
Time Frame: Immediately prior to first oral dose, up to 54 hours
Population: The Full Analysis Population for Efficacy consisted of subjects who received at least 1 dose of oral hydromorphone HCl and had at least 1 subsequent efficacy evaluation (pain measurement or supplemental pain medication).
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Oral ≥ 28 Days to < 13 Months: Infant and toddler - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- Oral ≥ 13 Months to < 5 Years: Young child - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- Oral ≥ 5 Years to < 12 Years: Older child - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
- Oral ≥ 12 Years to < 17 Years: Adolescent (Data for this group not collected. Test not appropriate for this age)
Arm/Group | Oral ≥ 28 Days to < 13 Months | Oral ≥ 13 Months to < 5 Years | Oral ≥ 5 Years to < 12 Years | Oral ≥ 12 Years to < 17 Years
Number analyzed (Participants) | 33 | 21 | 26 | 0
units on a scale
  Predose | 1.34 (0.388) | 2.67 (0.558) | 2.71 (0.522) |
  Dose 1 (1 hour postdose) | 1.13 (0.335) | 1.07 (0.483) | 2.17 (0.872) |
  Dose 2 (1 hour postdose) | 0.57 (0.223) | 0.67 (0.333) | 1.20 (0.583) |
  Dose 3 (1 hour postdose) | 0.27 (0.117) | 0.93 (0.715) | 0.75 (0.750) |
  Dose 4 (1 hour postdose) | 0.55 (0.274) | 0.85 (0.608) | 0.40 (0.400) |
  Dose 5 (1 hour postdose) | 0.70 (0.333) | 0.09 (0.091) | 1.00 (0.577) |
  Dose 6 (1 hour postdose) | 0.61 (0.465) | 1.20 (0.854) | 0.75 (0.479) |

3. Secondary Outcome: Mean (SE) of Faces Pain Scale-Revised (FPS-R) [Ages >= 5 Years-< 12 Years] Pain Scores on Hydromorphone Alone (Oral/Supplemental)Over Time
Description: Faces Pain Scale-Revised (FPS-R) consists of 6 facial expressions. Each face is 25 x 35 mm with 13 mm between faces. Each subject was asked to point to the face that reflected his or her pain. The end points are 0 = no pain and 10 = very much pain. The FPS-R scale was used for children over the age of 5 up to 12 years who have appropriate verbal skills.
Time Frame: Immediately prior to first oral dose with potentially up to 54 hours duration.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Oral ≥ 28 Days to < 13 Months: Infant and toddler (Data for this group not collected. Test not appropriate for this age)
- Oral ≥ 5 Years to <12 Years: Older child - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
Arm/Group | Oral ≥ 28 Days to < 13 Months | Oral ≥ 13 Months to < 5 Years | Oral ≥ 5 Years to <12 Years | Oral ≥ 12 Years to < 17 Years
Number analyzed (Participants) | 0 | 21 | 26 | 0
units on a scale
  Predose |  | 1.50 (0.957) | 2.59 (0.446) |
  Dose 1 (1 hour postdose) |  | 1.20 (1.200) | 2.25 (0.772) |
  Dose 2 (1 hour postdose) |  | 1.33 (1.333) | 0.92 (0.431) |
  Dose 3 (1 hour postdose) |  | 2.67 (0.667) | 1.54 (0.514) |
  Dose 4 (1 hour postdose) |  | 0 (0) | 1.86 (0.710) |
  Dose 5 (1 hour postdose) |  | 0 (0) | 1.64 (0.845) |
  Dose 6 (1 hour postdose) |  | 0 (0) | 0.40 (0.400) |

4. Secondary Outcome: Mean (SE) of Visual Analog Scale (VAS) [Ages 12-16] Pain Scores on Hydromorphone Alone (Oral/Supplemental) Over Time
Description: The Visual Analog Scale (VAS), a 10-cm Color Analog Scale anchored by the descriptors of 0 = "no pain" and 10 = "most pain," was used by children ≥ 12 years of age.
Time Frame: Immediately prior to first oral dose, up to 54 hours
Population: as for outcome 2
Measure: Mean (Standard Error); unit: unit on a scale
Groups:
- Oral ≥ 13 Months to < 5 Years: Young child (Data for this group not collected. Test not appropriate for this age)
- Oral ≥ 5 Years to <12 Years: Older child (Data for this group not collected. Test not appropriate for this age)
- Oral ≥ 12 Years to < 17 Years: Adolescent - received oral hydromorphone HCl every 6 hours, for a total of up to 9 doses, according to the dosing schedule. Starting doses were determined based on weight for this age group.
Arm/Group | Oral ≥ 28 Days to < 13 Months | Oral ≥ 13 Months to < 5 Years | Oral ≥ 5 Years to <12 Years | Oral ≥ 12 Years to < 17 Years
Number analyzed (Participants) | 0 | 0 | 0 | 20
unit on a scale
  Predose |  |  |  | 4.04 (0.530)
  Dose 1 (1 hour postdose) |  |  |  | 3.73 (0.629)
  Dose 2 (1 hour postdose) |  |  |  | 3.95 (0.673)
  Dose 3 (1 hour postdose) |  |  |  | 4.09 (0.569)
  Dose 4 (1 hour postdose) |  |  |  | 4.13 (0.599)
  Dose 5 (1 hour postdose) |  |  |  | 4.19 (0.945)
  Dose 6 (1 hour postdose) |  |  |  | 3.25 (0.998)

ADVERSE EVENTS:
Time Frame: AEs that were ongoing or were reported during the 7 days following the subject's last dose of study drug were followed until resolution or for 30 days. SAEs were followed until the event resolved or the sequelae stabilized.
Description: Adverse events were learned of through spontaneous reports and subject interview. The duration of treatment was up to 102 hours (up to 48 hours for the Parenteral Treatment Period and up to 54 hours for the Oral Treatment Period). Adverse events were collected for both parenteral and oral treatments.
Groups:
- Parenteral ≥ 28 Days to < 13 Months: Infant and toddler - received parenteral analgesia up to 48 hours postsurgery.
- Parenteral ≥ 13 Months to < 5 Years: Young child - received parenteral analgesia up to 48 hours postsurgery.
- Parenteral ≥ 5 Years to < 12 Years: Older child - received parenteral analgesia up to 48 hours postsurgery.
- Parenteral ≥ 12 Years to < 17 Years: Adolescent - received parenteral analgesia up to 48 hours postsurgery.
Arm/Group | Oral ≥ 28 Days to < 13 Months | Oral ≥ 13 Months to < 5 Years | Oral ≥ 5 Years to <12 Years | Oral ≥ 12 Years to < 17 Years | Parenteral ≥ 28 Days to < 13 Months | Parenteral ≥ 13 Months to < 5 Years | Parenteral ≥ 5 Years to < 12 Years | Parenteral ≥ 12 Years to < 17 Years
Serious Adverse Events (participants affected / at risk) | 2/39 | 2/23 | 1/29 | 0/25 | 3/39 | 0/23 | 1/29 | 1/25
Other Adverse Events (participants affected / at risk) | 21/39 | 14/23 | 15/29 | 6/25 | 27/39 | 16/23 | 19/29 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral ≥ 28 Days to < 13 Months (N=39) | Oral ≥ 13 Months to < 5 Years (N=23) | Oral ≥ 5 Years to <12 Years (N=29) | Oral ≥ 12 Years to < 17 Years (N=25) | Parenteral ≥ 28 Days to < 13 Months (N=39) | Parenteral ≥ 13 Months to < 5 Years (N=23) | Parenteral ≥ 5 Years to < 12 Years (N=29) | Parenteral ≥ 12 Years to < 17 Years (N=25)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion - DEATH (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Pre-treatment
Vascular procedure complication - DEATH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral ≥ 28 Days to < 13 Months (N=39) | Oral ≥ 13 Months to < 5 Years (N=23) | Oral ≥ 5 Years to <12 Years (N=29) | Oral ≥ 12 Years to < 17 Years (N=25) | Parenteral ≥ 28 Days to < 13 Months (N=39) | Parenteral ≥ 13 Months to < 5 Years (N=23) | Parenteral ≥ 5 Years to < 12 Years (N=29) | Parenteral ≥ 12 Years to < 17 Years (N=25)
Constipation (Gastrointestinal disorders) | 6 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 0 | 2 | 3 | 4
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 4 | 1 | 9 | 6 | 4 | 5
Sedation (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0 | 4 | 3 | 3 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1 | 2 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 1 | 2 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 0 | 2 | 5 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 1 | 10 | 5 | 6 | 8
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 11
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 5 | 3 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 11 | 4 | 2 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 8 | 3 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days